CLINICAL TRIAL: NCT03203434
Title: Non-invasive Detection of Anastomotic Leakage Following Esophageal and Pancreatic Surgery by Urinary Analysis
Brief Title: Non-invasive Detection of Anastomotic Leakage
Status: Completed | Type: Observational
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, Victor Plat, Principal investigator, Amsterdam UMC, location VUmc
Other Study IDs: 2014.543
Record Dates: First submitted 2017-06-27; First posted 2017-06-29 (Actual); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Anastomotic Leak
Keywords: Pancreatic cancer; Esophageal cancer; volatile organic compounds; Field asymmetric ion mobility spectrometry
MeSH Terms: conditions — Anastomotic Leak; Pancreatic Neoplasms; Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Biospecimen Retention: Samples Without DNA — Urine samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Esophageal anastomotic leakage
  Interventions: Diagnostic Test: Urinary volatile organic compound analysis
- Esophageal uncomplicated controls
  Interventions: Diagnostic Test: Urinary volatile organic compound analysis
- Pancreatic anastomotic leakage
  Interventions: Diagnostic Test: Urinary volatile organic compound analysis
- Pancreatic uncomplicated controls
  Interventions: Diagnostic Test: Urinary volatile organic compound analysis

INTERVENTIONS:
Diagnostic Test: Urinary volatile organic compound analysis

SUMMARY:
Esophagectomy or pancreaticoduodenectomy is the standard surgical approach for patients with malignant tumors of the esophagus or pancreatic head. These procedures are associated with high morbidity rates, which are strongly correlated with the occurrence of anastomotic leakage. Current diagnostic methods, including clinical, biochemical and radiological techniques are frequently inconclusive. Delay in diagnosis leads to delay in treatment, which ratifies the need for development of novel and accurate non-invasive diagnostic tests for detection of anastomotic leakage. Urinary volatile organic compounds reflect the metabolic status of an individual, which is associated with a systemic immunological response. The aim of this study was to determine the diagnostic accuracy of urinary volatile organic compounds to detect anastomotic leakage after esophagectomy or pancreaticoduodenectomy in an early phase.

ELIGIBILITY:
Inclusion Criteria:

* Patients were aged 18-90 years
* American Society of Anesthesiologists (ASA) physical status of 3 or lower
* All participants were capable to understand the study information and signed written informed consent

Exclusion Criteria:

* None

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible participants had suspected malignancies of the esophagus, pancreas, distal bile duct, ampulla Vateri or duodenum and were scheduled for surgery (i.e. esophagectomy or pancreaticoduodenectomy).
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2017-03-01 (Actual); Study Completion 2017-03-01 (Actual)

PRIMARY OUTCOMES:
Anastomotic leakage | Postoperatively (30-days)

CONTACTS AND LOCATIONS:
Overall Officials: Freek Daams, MD PhD, Study Director — Amsterdam UMC, location VUmc

IPD SHARING:
Plan to Share IPD: No